CLINICAL TRIAL: NCT04288154
Title: The Impact of Training With Whole Body-EMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 19-003449
Record Dates: First submitted 2020-01-24; First posted 2020-02-28 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EMS Group - Experimental (Experimental): EMS device will be turned on during exercise for this group.
  Interventions: Device: EMS Device On
- EMS Group - Control (Placebo Comparator): EMS device will be turned off during exercise for this group.
  Interventions: Other: EMS Device Off

INTERVENTIONS:
Device: EMS Device On — The EMS Device will turned on during exercise as opposed to it being turned off for control group.
  Arms: EMS Group - Experimental
Other: EMS Device Off — The EMS Device will turned off during exercise as opposed to it being turned off for control group.
  Arms: EMS Group - Control

SUMMARY:
Researchers are trying to find out what impact training with whole body-EMS (Electronic muscle stimulation) has on various health outcomes.

DETAILED DESCRIPTION:
All subjects in both groups who enroll into this study will undergo an assessment of peripheral endothelial function with reactive hyperemia-peripheral arterial tonometry (RH-PAT) testing using EndoPAT; an assessment of vital signs including heart rate, blood pressure, weight, height and body mass index; laboratory blood work; cardiorespiratory testing using treadmill testing to determine VO2 max and maximal tolerated heart rate; maximal strength and maximal power testing on chest press and leg press testing; and percent body fat and fat distribution testing at baseline, and at 16-weeks follow-up (immediately after completing a 16-week training program using whole body-EMS). Baseline cardiovascular risk factors will be assessed by subject questionnaire and verified by chart review. In addition, subjects will complete an angina/chest pain symptom questionnaire (Rose Questionnaire), quality of life questionnaire (LASA Questionnaire), depression questionnaire (Patient Health Questionaire-9) and perceived stress questionnaire (Perceived Stress Scale) to assess for psychosocial wellness at each point in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Employees at the Mayo Clinic, Rochester, MN

Exclusion Criteria:

* Subjects under the age of 18
* Pregnant women
* Subjects with a history of liver or kidney disease, acute illness, taking medications (such as glucocorticoids)
* Subjects who have conditions (such as chronic inflammatory muscular diseases or Cushing's syndrome) that affect muscle mass
* Individuals with pacemakers and implantable cardiac defibrillators
* Individuals who conduct any other type of resistance training (> 45 minutes/week)
* Individuals who have regular "high" alcohol consumption (> 80g/day on 5 days a week)
* Subjects unable to consent to or participate in the 16-week EMS intervention or be available for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Electro Muscle Stimulation (EMS) Group Experimental: EMS device was turned on during exercise for this group.
  EMS Device On: The EMS Device was turned on during exercise as opposed to it being turned off for control group.
- EMS Group - Control: EMS device was turned off during exercise for this group.
  EMS Device Off: The EMS Device was turned off during exercise as opposed to it being turned off for control group.
Period: Overall Study
Arm/Group | Electro Muscle Stimulation (EMS) Group Experimental | EMS Group - Control
Started | 46 | 32
Completed | 37 | 23
Not Completed | 9 | 9
Not completed — Withdrawal by Subject | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- EMS Group - Experimental: EMS device was turned on during exercise for this group.
  EMS Device On: The EMS Device was turned on during exercise as opposed to it being turned off for control group.
- Total: Total of all reporting groups
Arm/Group | EMS Group - Experimental | EMS Group - Control | Total
Number analyzed (Participants) | 46 | 32 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.8) | 35.6 (9.7) | 35.65 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 19 | 47
  Male | 18 | 13 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 46 | 32 | 78

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Reactive Hyperemia Index (RHI)
Description: Mean change in RHI. RHI measured by noninvasive endothelial peripheral arterial tomography (EndoPat) test. The EndoPAT involves probes on the index fingers of both hands & evaluating the blood flow to one hand before & after inflating a blood pressure (BP) cuff on one arm, temporarily reducing blood flow to the fingers. The finger sensor on the affected arm will show no blood flow, the sensor on the opposite index finger will display normal blood flow level. After several minutes, the BP cuff is released, allowing blood to flow back into the affected lower arm. If the finger sensor on the affected arm shows a rush of blood, the blood vessels are functioning normally. If the blood flow return is sluggish, the blood vessels are unhealthy. EndoPAT results are reported as the "Endoscore" (range 0-3); a score of 1.67 and lower indicates the need for immediate medical attention; a score between 1.68 and 2 indicates a need to reduce risk factors; a score above 2.1 indicates a healthy heart.
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
score on a scale | 0.02 (0.1) | -0.26 (0.3)

2. Secondary Outcome: Change in BMI
Description: Subject's BMI calculated as weight in kilograms divided by height in meters squared. Uses measurements of height and weight obtained during study (with appropriate metric conversions)
Time Frame: baseline,16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 46 | 32
kg/m^2 | 0.2 (0.9) | 0.06 (0.5)

3. Secondary Outcome: Change in Total Cholesterol
Description: Total cholesterol is the sum of a person's HDL cholesterol, LDL cholesterol, and 20% of their triglyceride levels. Healthy total cholesterol is less than 200 mg/dL of blood
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
mg/dL | -1.7 (25.1) | 19.2 (26.5)

4. Secondary Outcome: Change in Maximal Oxygen Consumption (VO2max)
Description: VO2 max, or maximal oxygen consumption, refers to the maximum amount of oxygen that an individual can utilize during intense or maximal exercise. VO2 max is the number of milliliters of oxygen used per kilogram of body weight in one minute (ml/kg/min)
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
ml/kg/min | 0.3 (3.4) | 1.1 (3.9)

5. Secondary Outcome: Mean Change in Quality-of-Life Score as Measured by the Longitudinal Amsterdam Aging Study (LASA) Questionnaire:
Description: The LASA is subject reported ten item quality of life questionnaire. The ten items are scored from 0 -10, 0 being as bad as it can be and 10 being as good as it can be. Total scores range from 0 - 100, lower scores indicate being as bad as it can be, higher scores indicate being as good as it can be.
Time Frame: baseline, week 16
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
score on a scale | 0.04 (0.9) | 0.3 (0.5)

6. Secondary Outcome: Change in Creatinine Kinase (CK)
Description: A creatine kinase test may be used to detect inflammation of muscles or muscle damage due to muscle disorders. A person may have muscle injury with few or nonspecific symptoms, such as weakness, fever, and nausea, that may also be seen with a variety of other conditions. A healthcare practitioner may use a CK test to help detect muscle damage in these cases, especially if someone is taking a drug such as a statin. Normal values at rest are usually between 60 and 174 U/L.
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
U/L | 417.9 (1499) | -137.2 (375.9)

7. Secondary Outcome: Mean Change in Stress Score as Measured by the Perceived Stress Scale
Description: The Perceived Stress Scale is a subject reported 10 item stress questionnaire. The 10 items are scored from 0 to 4, with 0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often and 4 = very often. Total scores range from 0 - 40, lower scores indicate lower stress, and higher scores indicate higher stress.
Time Frame: baseline, week 16
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
score on a scale | -1.0 (5.5) | -0.4 (4.8)

8. Secondary Outcome: Mean Change in Depression Score as Measured by the Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 Screens for the presence and severity of depression with 9 questions in a scale of 0-3. Zero=not at all, 1=several days, 2=more than half the days, 3=nearly every day. Total scores range 0 - 27. A total score of 0-4=minimal depression, 5-9=mild depression, 10-14=moderate depression, 15-19=moderately severe depression, 20-27=severe depression
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
score on a scale | -0.3 (3.2) | 0.05 (1.2)

9. Secondary Outcome: Change in Blood Glucose
Description: Sugar in the form of glucose in the blood. The concentration of glucose in the blood. A healthy normal range is 70 to 99 mg/dL
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
mg/dL | 0.7 (10.3) | -0.8 (8.8)

10. Secondary Outcome: Change in HbA1c
Description: Hemoglobin is a protein within red blood cells. As glucose enters the bloodstream, it binds to hemoglobin, or glycates. The more glucose that enters the bloodstream, the higher the amount of glycated hemoglobin. An A1C level below 5.7 percent is considered normal. Reported as percentage of glycated hemoglobin
Time Frame: baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
percentage of glycated hemoglobin | -0.01 (0.2) | 0 (0.2)

11. Secondary Outcome: Change in High Sensitivity C- Reactive Protein (CRP)
Description: High sensitivity C-reactive protein is a substance produced by the liver in response to inflammation. Normal CRP levels are below 3.0 mg/L
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
mg/L | 0.06 (0.7) | 0.3 (2.3)

12. Secondary Outcome: Change in Uric Acid:
Description: Uric acid is a heterocyclic compound of carbon, nitrogen, oxygen, and hydrogen. Uric acid is a product of the metabolic breakdown of purine nucleotides. Normal blood values are 1.5 to 6.0 milligrams/deciliter (mg/dL) for women and 2.5 to 7.0 mg/dL for men
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
mg/dL | 0.1 (0.6) | 0.2 (0.6)

13. Secondary Outcome: Change in Fibrinogen
Description: Fibrinogen is a protein produced by the liver. This protein helps stop bleeding by helping blood clots to form. Blood fibrinogen is the amount of fibrinogen in a blood sample. Normal range is 200 to 400 mg/dL
Time Frame: Baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
mg/dL | 5.4 (27.3) | 9.0 (34.8)

14. Secondary Outcome: Change in Homocysteine
Description: Homocysteine is an amino acid which occurs in the body as an intermediate in the metabolism of methionine and cysteine. Normal range 4 and 15 micromoles/liter (µmol/L)
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
µmol/L | -6.7 (32.8) | -0.7 (32.8)

15. Secondary Outcome: Change in Lipoprotein
Description: Lipoprotein is a type of protein that combine with and transport fat or other lipids in the blood plasma. Normal range is less than 30 mg/dL
Time Frame: baseline, 16 weeks
Population: Data was not collected or analyzed for 9 subjects in each arm
Measure: Mean (Standard Deviation); unit: 30 mg/dL
Arm/Group | EMS Group - Experimental | EMS Group - Control
Number analyzed (Participants) | 37 | 23
30 mg/dL | 5.6 (20.9) | 15.4 (38.0)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 16 weeks
Arm/Group | EMS Group - Experimental | EMS Group - Control
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/32
Other Adverse Events (participants affected / at risk) | 0/46 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT04288154/Prot_SAP_000.pdf